CLINICAL TRIAL: NCT06449014
Title: Efficacy of Mini-Implant-Assisted Maxillary Expansion on Late Adolescents and Adults and Its Effects on Nasal Permeability and Airway Volume Using Three Different Activation Protocols: A Randomized Controlled Trial (MARPE_1)
Brief Title: Efficacy of Mini-implant Assisted Maxillary Expansion in Adolescents and Adults
Acronym: MARPE_1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Erasme_MARPE_1
Record Dates: First submitted 2024-05-23; First posted 2024-06-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-12

CONDITIONS: Narrow Maxilla
Keywords: MARPE; Endognathia; rhinomanometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRAP (Experimental): Continuous Rapid Activation Protocol: 1 activation of the expansion screw per day which is equal to 0,17 mm expansion of the maxilla per day till reaching the clinical goal
  Interventions: Device: Mini-implants assisted maxillary expansion
- SCAP (Experimental): Continuous Slow Activation Protocol: 2 activations of the expansion screw which is equal to 0,33 mm expansion of the maxilla per day during the first 7 days. After that first week, then each third day 1 activation (0,17 mm / 3 days).
  Interventions: Device: Mini-implants assisted maxillary expansion
- FCPC (Experimental): force-controlled polycyclic protocol: 2 activations of the expansion screw which is equal to 0,33 mm expansion of the maxilla per day during the first 7 days. Then the expansion screw will be turned 6 sides backward, and after 15 min, the expansion screw will be turned forward 6 sides again. And every third day, the device will be additionally activated by 0.17mm (0,17 mm / 3 days)
  Interventions: Device: Mini-implants assisted maxillary expansion

INTERVENTIONS:
Device: Mini-implants assisted maxillary expansion — The intervention involved the placement of orthodontic mini-screws in the patient's palate, varying in diameter from 2 to 2.3 mm and in length from 11 to 15 mm. After mini-screw insertion, another intraoral scan was taken for the fabrication of the appliance. Approximately three weeks later, the expander was placed in the patient's palate, and maxillary expansion was initiated immediately afterward according to the chosen protocol.
  Other Names: Mini-screws assisted maxillary expansion; Mini-implants assisted rapid maxillary expansion

SUMMARY:
Transverse maxillary deficiency is a common orthodontic issue, affecting around 10% of adults. Late adolescents and adults often require more force to expand the midpalatal suture due to its increased interdigitation. This study aims to assess the effectiveness of MARPE in this demographic and determine the best activation protocol for non-surgical maxillary expansion using mini-screw-supported appliances. Additionally, the study will evaluate the effectiveness of MARPE on nasal permeability and airway volume.

DETAILED DESCRIPTION:
The study design comprised a three-arm, parallel-group randomized controlled trial (RCT) conducted at the Orthodontics clinic of Brussels University Hospital. Patients were randomly allocated into one of three groups:

1. Continuous rapid activation protocol: Patients received one activation of 0.17 mm per day until reaching the clinical goal.
2. Continuous slow activation protocol: Patients underwent two activations (0.33 mm) per day for the first 7 days, followed by one turn forward every third day (0.17 mm / 3 days).
3. Force-controlled polycyclic protocol: Patients underwent two activations (0.33 mm) per day for the first 7 days. Then, the hex nut was turned 6 sides backward, followed by 6 sides forward after 15 minutes. Additionally, the device was activated by 0.17 mm every third day.

Intervention:

All patients underwent maxillary expansion with MARPE. Four orthodontic mini-screws were inserted under local anesthesia using a surgical guide and motor. Surgical incision was not required, and predrilling was performed if necessary. The MARPE remained in place for 12 months after expansion to allow bone remodeling in the midpalatal suture. Fixed straight-wire treatment commenced 2 months after expansion termination. Patients underwent retention check-ups at 6 and 12 months post-expansion, and expansion screws and mini-screws were removed after 12 months or before orthognathic surgery, if applicable.

The specific aims of the study were to evaluate the success rate of nonsurgical maxillary expansion, compare the efficacy of the three activation protocols, assess and compare complications, analyze the correlation between success rate and Midpalatal Suture Maturation Stage (MPS), age, and sex, and measure nasal permeability variation using anterior rhinomanometry.

ELIGIBILITY:
Inclusion Criteria:

* from the age of 16 onwards
* who presented with transverse maxillary discrepancy (unilateral, bilateral, anticipated, or constriction without crossbite).

Exclusion Criteria:

* history or presence of maxillofacial surgery, cleft lip and palate, craniofacial anomalies or syndromes, congenital tooth anomalies, and periodontal disease.
* Patients who had previously palatal expansion were excluded also.
* Presence of anatomic or pathological obstacle of the palatal mini-screw insertion (impacted tooth, tumor.)
* refusal of study participation

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
MPSM: mid-palatal suture middle molars | up to 6 months
  the width of the mid-palatal suture measure in millimeters at the level of the first molars
ANS-ANS | up to 6 months
  the distance in millimeters between the right anterior nasal spine and the left anterior nasal spine after the maxillary expansion
PNS-PNS | up to 6 months
  distance in millimeters between the right posterior nasal spine and the left posterior nasal spine after the maxillary expansion
UID | up to 6 months
  distance in millimeters from the most external point of the right frontozygomatic suture to the most external point of the left frontozygomatic suture.
ZMA | up to 6 months
  width in millimeters between the right and left zygomatic arches at its widest point at the most inferior level of the orbits.
LID: | up to 6 months
  distance in millimeters from the most external point of the right zygomaticomaxillary suture to the most external point of the left zygomaticomaxillary suture
NCW: nasal cavity width | up to 6 months
  Transverse distance in millimeters between the left and right most lateral point of the nasal cavity
MSW: midpalatal suture width | up to 6 months
  Transverse distance in millimeters between the medial limits of the left and right palatal process at the palatal floor
IMW: intermolar width | up to 6 months
  Transverse distance in millimeters between the left and right maxillary M1 mesiocentral fossae
IPW: interpremolar width | up to 6 months
  Transverse distance in millimeters between the left and right maxillary P1 mesial fossae
ICW: intercanine width | up to 6 months
  Transverse distance in millimeters between the left and right maxillary canine buccal cusp tips
PAW: palatal alveolar width | up to 6 months
  Transverse distance between in millimeters the left and right most cervical medial limits of the palatal alveolar process
TI : tooth inclination | up to 6 months
  2D inner angle (in degrees) between the palatal plane and the left and right line running through the palatal apex and the mesiobuccal fossa or the mesial fossa

SECONDARY OUTCOMES:
RT resistance total | up to 6 months
  Total bilateral nasal resistance in Pa.s.cm³
NCV: nasal cavity volume | up to 6 months
  nasal cavity volume in mm3
RMSV : right maxillary sinus volume | up to 6 months
  Right maxillary sinus volume in mm3
LMSV : left maxillary sinus volume | up to 6 months
  left maxillary sinus volume in mm3
NPV nasopharynx volume | up to 6 months
  nasopharynx volume in mm3
OPV oropharynx volume | up to 6 months
  OPV oropharynx volume in mm3
OMCSA: oropharynx minimum cross-sectional area | up to 6 months
  oropharynx minimum cross-sectional area in mm2
AV: Accumulated volume | up to 6 months
  which represents the total volume in mm3, is calculated using the sum of the NCV, RMSV, LMSV, NPV, and OPV

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Route de Lennik 900, Anderlecht, Brussels Capital
  - service dentaire et d'orthodontie de l'hopital université de bruxelles (HUB), Anderlecht, Brussels Capital